CLINICAL TRIAL: NCT01462526
Title: The Detection of Glaucoma Using Pupillography
Acronym: RAPiD
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00044899
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Participants who do not have glaucoma in either eye
- Glaucoma: Participants who have glaucoma in one or both eyes

SUMMARY:
Current screening methods for glaucoma detection are not perfect and nearly half of those in the United States with glaucoma go undiagnosed. Minority populations are even less likely to be diagnosed. Better screening methods are needed to identify the undiagnosed and to provide them care that can help them retain good vision.

Glaucoma is often more severe in one eye and this fact can be exploited in screening tests. The investigators plan to use a novel screening device that very accurately records the pupillary response from each eye. It is likely that patients with glaucoma will have abnormal responses when measured, and by comparing responses between the two eyes the investigators will be able to determine who has glaucoma. If this test works well, it will provide a low-cost way to screen populations at risk for glaucoma. Furthermore, this research will expand the knowledge base regarding how pupil responses to light differ between persons with and without glaucoma. Insights gained from this study will be useful in the development of an effective screening tool in the detection of glaucoma.

DETAILED DESCRIPTION:
Glaucoma is often asymmetric in nature, and an afferent pupillary defect (APD) is frequently present in persons with glaucoma. The investigators propose to conduct a clinic-based prospective study to assess the accuracy of using a binocular pupillographic device (RAPiD, Konan Medical, USA) to detect people with glaucoma. This device is designed to record and analyze pupil responses at multiple, controlled stimulus intensities, while using varied patterns and color stimuli.

The asymmetric nature of glaucoma suggests that a high proportion of persons with glaucoma will have an APD (although many may be subtle and would be missed with less refined testing methods). When glaucoma patients have severe nerve damage or when field loss is bilateral and symmetric, an APD may not be present or may be too small to detect. Noting this limitation, the investigators will compare pupillary responses to stimuli at different locations (for example the superior compared to the inferior hemifield) to determine whether the investigators can detect asymmetric glaucoma damage within the same eye. In addition, it is likely that the pupil response in glaucoma will be diminished when compared to normal, which will also help with detection.

Aim1: To examine the amplitude, latency and velocity of the pupil light reflex by optimizing its measurement to stimuli of various intensities and colors, and to characterize the variability of this response in normal subjects.

Aim2: To quantify the amount of structural loss (retinal nerve fiber layer thickness and optic nerve head parameters) and functional loss (visual field mean deviation) necessary for an APD (as detected by RAPiD) to manifest.

Aim3a: To develop an algorithm that best discriminates those with and without glaucoma by individual or combined use of 1) detecting an APD between the two eyes, 2) comparing pupil responses in different parts of the visual field within the same eye, and 3) comparing responses of diseased eyes to responses of "normal" eyes.

Aim 3b: To assess the validity of this algorithm in glaucoma detection and to assess the reproducibility of the pupil response measurements at a follow-up visit within 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older at enrollment
* Presenting visual acuity better than 20/100 in both eyes
* Spherical equivalent refractive error within the range of 4.0 and -6.0 diopters in both eyes

Exclusion Criteria:

* Ocular surgery in either eye within 3 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with glaucoma, glaucoma suspects, or ocular hypertension who present to the glaucoma service at the Johns Hopkins Wilmer Eye Institute. We will also recruit normal subjects from the accompanying persons of patients attending examinations who are not blood relatives of the patient.
Sampling Method: Non-Probability Sample
Enrollment: 798 (Actual)
Dates: Start 2011-03; Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Friedman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute Johns Hopkins University, Baltimore, Maryland, United States